CLINICAL TRIAL: NCT02922153
Title: The cryoICE™ CryoAnalgesia Study For Pain Management in Post thoRacic Procedures Via intercOSTal Cryoanalgesia (FROST)
Acronym: FROST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP2015-4
Record Dates: First submitted 2016-09-26; First posted 2016-10-04 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-04

CONDITIONS: Pain
Keywords: CryoAnalgesia; Thoracotomy; Forced Expiratory Volume (FEV1); Visual Analog Scale (VAS)
MeSH Terms: conditions — Pain | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cryoanalgesia + Standard of Care (SOC) (Experimental): Cryoanalgesia in Conjunction with Standard of Care. Up to 5 sessions of cryoanalgesia for 120 seconds per session.
  Interventions: Device: Cryoanalgesia; Drug: Standard of Care
- Standard of Care (Active Comparator): Institutional SOC for pain management will be followed. The use of local post-operative pain management techniques (i.e., intercostal, peri-vertebral, or any other acceptable method) is permitted for both treatment groups up to 24 hours post-operatively according to institutional standard of care.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Device: Cryoanalgesia — AtriCure® cryoICE cryo-ablation system
  Other Names: cryoICE
  Arms: Cryoanalgesia + Standard of Care (SOC)
Drug: Standard of Care — Institutional SOC for pain management will be followed.
  Other Names: SOC

SUMMARY:
The investigators propose to assess whether intra-operative intercostal cryoanalgesia using the cryoICE® probe (AtriCure®, Inc., 7555 Innovation Way, Mason, Ohio) provides superior post-operative analgesic efficacy as compared to current pain management in patients undergoing unilateral thoracotomy cardiac procedures.

DETAILED DESCRIPTION:
Completion of the proposed study will for the first time demonstrate efficacy of intercostal cryoanalgesia in patients undergoing minimally invasive cardiac procedures. Furthermore, results of this study may have a pivotal role in supporting future clinical outcome trials for intercostal cryoanalgesia therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 85 years male or female
* Patients undergoing unilateral thoracotomy cardiac procedures (with the exception of Aortic Aneurysm repair as sole treatment)
* Acceptable surgical candidate, including use of general anesthesia
* Willing and able to provide written informed consent
* Willing and able to return for scheduled follow-up visits

Exclusion Criteria:

* Cardiac valve surgical procedure via conventional full sternotomy
* Procedures that require a posterolateral thoracotomy
* Current pregnancy
* Current use of prescription opioids
* FEV1 < 40% predicted
* Documented myocardial infarction within 30 days of signing Informed Consent Form (ICF)
* Documented psychiatric disease
* Documented chronic pain syndrome
* Documented history of substance abuse
* Patient currently enrolled in another research study that could directly affect results of either study
* Physical or mental condition that would interfere with patient's self-assessment of pain
* Disqualifying medical condition per investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lau, MD, Principal Investigator — Corewell Health East
Locations (5):
- United States (5):
  - University of Southern California (USC), Los Angeles, California
  - University of Michigan, Ann Arbor, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - United Heart and Vascular Institute - Allina, Saint Paul, Minnesota
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sepsas E, Misthos P, Anagnostopulu M, Toparlaki O, Voyagis G, Kakaris S. The role of intercostal cryoanalgesia in post-thoracotomy analgesia. Interact Cardiovasc Thorac Surg. 2013 Jun;16(6):814-8. doi: 10.1093/icvts/ivs516. Epub 2013 Feb 19. PMID 23424242
- [Background] Moorjani N, Zhao F, Tian Y, Liang C, Kaluba J, Maiwand MO. Effects of cryoanalgesia on post-thoracotomy pain and on the structure of intercostal nerves: a human prospective randomized trial and a histological study. Eur J Cardiothorac Surg. 2001 Sep;20(3):502-7. doi: 10.1016/s1010-7940(01)00815-6. PMID 11509270
- [Background] Glauber M, Karimov JH, Farneti PA, Cerillo AG, Santarelli F, Ferrarini M, Del Sarto P, Murzi M, Solinas M. Minimally invasive mitral valve surgery via right minithoracotomy. Multimed Man Cardiothorac Surg. 2009 Jan 1;2009(122):mmcts.2008.003350. doi: 10.1510/mmcts.2008.003350. PMID 24415737
- [Background] Loan WB, Dundee JW. The clinical assessment of pain. Practitioner. 1967 Jun;198(188):759-68. No abstract available. PMID 4859864
- [Background] PAPPER EM, BRODIE BB, ROVENSTINE EA. Postoperative pain; its use in the comparative evaluation of analgesics. Surgery. 1952 Jul;32(1):107-9. No abstract available. PMID 14950594
- [Background] Katz J. Cryoanalgesia for postthoracotomy pain. Ann Thorac Surg. 1989 Jul;48(1):5. doi: 10.1016/0003-4975(89)90166-5. No abstract available. PMID 2764599
- [Background] Cook TM, Riley RH. Analgesia following thoracotomy: a survey of Australian practice. Anaesth Intensive Care. 1997 Oct;25(5):520-4. PMID 9352765
- [Background] SIMPSON BR, PARKHOUSE J, MARSHALL R, LAMBRECHTS W. Extradural analgesia and the prevention of postoperative respiratory complications. Br J Anaesth. 1961 Dec;33:628-41. doi: 10.1093/bja/33.12.628. No abstract available. PMID 13913200
- [Background] Maiwand MO, Makey AR, Rees A. Cryoanalgesia after thoracotomy. Improvement of technique and review of 600 cases. J Thorac Cardiovasc Surg. 1986 Aug;92(2):291-5. PMID 3736085
- [Background] Gough JD, Williams AB, Vaughan RS, Khalil JF, Butchart EG. The control of post-thoracotomy pain. A comparative evaluation of thoracic epidural fentanyl infusions and cryo-analgesia. Anaesthesia. 1988 Sep;43(9):780-3. doi: 10.1111/j.1365-2044.1988.tb05757.x. PMID 3255292
- [Background] Gwak MS, Yang M, Hahm TS, Cho HS, Cho CH, Song JG. Effect of cryoanalgesia combined with intravenous continuous analgesia in thoracotomy patients. J Korean Med Sci. 2004 Feb;19(1):74-8. doi: 10.3346/jkms.2004.19.1.74. PMID 14966345
- [Derived] Lau WC, Shannon FL, Bolling SF, Romano MA, Sakwa MP, Trescot A, Shi L, Johnson RL, Starnes VA, Grehan JF. Intercostal Cryo Nerve Block in Minimally Invasive Cardiac Surgery: The Prospective Randomized FROST Trial. Pain Ther. 2021 Dec;10(2):1579-1592. doi: 10.1007/s40122-021-00318-0. Epub 2021 Sep 20. PMID 34545530

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cryoanalgesia + Standard of Care (SOC) | Standard of Care
Started | 65 | 19
Completed | 55 | 17
Not Completed | 10 | 2
Not completed — Death | 8 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cryoanalgesia + Standard of Care (SOC) | Standard of Care | Total
Number analyzed (Participants) | 65 | 19 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.83 (11.96) | 66.42 (12.53) | 64.42 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 8 | 35
  Male | 38 | 11 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 59 | 18 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 65 | 19 | 84
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.61 (5.03) | 29.95 (4.73) | 28.91 (4.96)
Forced Expiratory Value (FEV1) [Mean (Standard Deviation); unit: Liters (L)] | 2.33 (0.78) | 2.28 (0.84) | 2.32 (0.79)
Visual Analog Scale (general) [Mean (Standard Deviation); unit: units on a scale] — 0-10 Numeric Pain Rating Scale
  units on a scale | 0.32 (0.95) | 0.42 (0.90) | 0.35 (0.94)
Visual Analog Scale (surgical site) [Mean (Standard Deviation); unit: units on a scale] — 0-10 Numeric Pain Rating Scale at the surgical site.
  units on a scale | 0.03 (0.25) | 0.21 (0.54) | 0.07 (0.34)
Society of Thoracic Surgeon Score (STS) [Mean (Standard Deviation); unit: Percentage] — Risk of Mortality Percentage - High is greater than or equal to 8%, intermediate is greater than or equal to 4% and low is less than 4%. Population: The information required in this data field was not obtained on five of the sixty-five participants. Data was reported on sixty participants.
  Percentage
    number analyzed (Participants) | 60 | 19 | 79
    (all) | 2.03 (1.90) | 2.86 (2.57) | 2.23 (2.09)

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome 1: Forced Expiratory Volume (FEV1) at 48-Hours Post-Surgery
Description: Forced Expiratory Volume (FEV1) is the measurement of how much air, in volume, that a person can exhale with a forced breath. It is measured using a spirometer device.
Time Frame: 48-hours post-surgery
Population: Includes all patients who were consented and randomized (84). Not all subjects in each of the arms participated. Some refused to participate or were unable to participate in data collection which resulted in fewer subjects able to be analyze. This resulted in 46/64 subject for Cryoanalgesia (CRYO) + SOC and 16/19 subjects for SOC.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters (L)
Groups:
- Cryoanalgesia + SOC: Cryoanalgesia in Conjunction with Standard of Care. Up to 5 sessions of cryoanalgesia for 120 seconds per session.
  Cryoanalgesia: AtriCure® cryoICE cryo-ablation system
  Standard of Care: Institutional SOC for pain management will be followed.
Arm/Group | Cryoanalgesia + SOC | Standard of Care
Number analyzed (Participants) | 46 | 16
Liters (L) | 1.2 [1.10 to 1.31] | 0.93 [.71 to 1.14]
Statistical Analysis 1: Comparison: Cryoanalgesia + SOC vs Standard of Care; Test type: Superiority; p = 0.0223, t-test, 1 sided; One-sided, two-sample t-test

2. Primary Outcome: Primary Outcome 2: Visual Analogue Scale (VAS) Pain in the Surgical Region at 48-Hours Post-Surgery
Description: The Visual Analogue Scale (VAS) uses a picture of a linear scale that shows numbers 0-10 with 0 being the least amount of pain and 10 being the most amount of pain. This outcome looked at pain in the surgical region specifically.
Time Frame: 48-hours post-surgery
Population: Analysis population includes all patients who were consented and randomized (84). However, not all subjects in each of the arms participated. Some refused to participate or were unable to participate in data collection which resulted in fewer subjects able to be analyze. This resulted in 61/64 subject for CRYO + SOC and 18/19 subjects for SOC.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cryoanalgesia + SOC | Standard of Care
Number analyzed (Participants) | 61 | 18
units on a scale | 2.82 (2.70) | 3.06 (2.82)
Statistical Analysis 1: Comparison: Cryoanalgesia + SOC vs Standard of Care; Test type: Superiority; p = 0.6259, t-test, 1 sided; One-sided two-sample t-test
Statistical Analysis 2: Comparison: Cryoanalgesia + SOC vs Standard of Care; Test type: Superiority; p = 0.518, Wilcoxon (Mann-Whitney); Wilcoxon two-sample test

3. Secondary Outcome: Secondary Outcome 1: Spirometry Assessments at 48-Hours Post-Extubation
Description: Spirometry assessments measured included: forced expiratory volume (FEV1), forced vital capacity (FVC) and slow vital capacity (SVC), all of which are measured with a spirometer. FEV1 is the amount of air forcibly expired during the first second of breath, FVC is the total volume of air expired over the whole forced breath and SVC is the total volume over the whole breath but at a slow pace, not forced.
Time Frame: 48-hours post-extubation
Population: Analysis population includes all patients who were consented and randomized (84). However, not all subjects in each of the arms participated. Some refused to participate or were unable to participate in data collection which resulted in fewer subjects able to be analyze. This resulted in 46/64 subject for CRYO + SOC and 16/19 subjects for SOC.
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Cryoanalgesia + SOC | Standard of Care
Number analyzed (Participants) | 46 | 16
Liters (L)
  FEV1 | 1.20 (0.46) | 0.93 (0.43)
  FVC | 1.60 (0.62) | 1.33 (0.55)
  SVC | 1.52 (0.61) | 1.28 (0.55)
Statistical Analysis 1: Comparison: Cryoanalgesia + SOC vs Standard of Care; Test type: Superiority; p = 0.0201, t-test, 1 sided — FEV1 one-sided, two-sample t-test
Statistical Analysis 2: Comparison: Cryoanalgesia + SOC vs Standard of Care; Test type: Superiority; p = 0.06, t-test, 1 sided — FVC one-sided, two-sample t-test
Statistical Analysis 3: Comparison: Cryoanalgesia + SOC vs Standard of Care; Test type: Superiority; p = 0.09, t-test, 1 sided — SVC one-sided, two-sample t-test

4. Secondary Outcome: Secondary Outcome 2: Visual Analogue Scale (VAS) Pain at the 72, 96 and 120-Hours Post-Op Time Points
Description: as for outcome 2
Time Frame: 72-, 96- and 120-hours Post-Op
Population: Number of participants decreases at each subsequent visit due to patients being discharged at different time points during hospital stay.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cryoanalgesia + SOC | Standard of Care
Number analyzed (Participants) | 64 | 19
units on a scale
  72 Hours Post-Op: number analyzed (Participants) | 59 | 18
  72 Hours Post-Op | 2.08 (2.39) | 1.44 (2.09)
  96 Hours Post-Op: number analyzed (Participants) | 51 | 15
  96 Hours Post-Op | 1.84 (2.39) | 2.00 (2.45)
  120 Hours Post-Op: number analyzed (Participants) | 42 | 10
  120 Hours Post-Op | 2.50 (2.82) | 2.40 (3.37)
Statistical Analysis 1: Comparison: Cryoanalgesia + SOC vs Standard of Care; Test type: Superiority; p = 0.3085, Wilcoxon (Mann-Whitney) — 72 Hours Post-Op; Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Cryoanalgesia + SOC vs Standard of Care; Test type: Superiority; p = 0.8196, Wilcoxon (Mann-Whitney) — 96 Hours Post-Op; Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Cryoanalgesia + SOC vs Standard of Care; Test type: Superiority; p = 0.7269, Wilcoxon (Mann-Whitney) — 120 Hours Post-Op; Wilcoxon rank-sum test

5. Secondary Outcome: Secondary Outcome 3: Allodynia at the 3 and 6 Month Visit
Description: Allodynia is pain around surgical site. It is pain that occurs from stimuli that are not normally painful such as a light touch or a brush of hair around where the surgery took place.
Time Frame: 3 and 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoanalgesia + SOC | Standard of Care
Number analyzed (Participants) | 64 | 19
Participants
  3 Month | 0 | 0
  6 Month | 1 | 0

6. Secondary Outcome: Secondary Outcome 4: Duration of Oral Endotracheal Intubation From Extubation Until the Patient Leaves the Operating Room
Description: Oral endotracheal intubation is where a patient has a tube placed down their throat and into the trachea, the large airway from the mouth to the lungs. This is done to ensure that patients who are asleep under anesthesia are able to fully breath. This outcome measured the hours from the time the patient leaves the operating room until they were extubated, or had the tube removed from their trachea.
Time Frame: Hours until patient is extubated from time patient leaves the operating room
Population: Overall number is for all patients that were fully extubated and accounts for patients who were unable to be extubated or did were unable to finish extubation.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cryoanalgesia + SOC | Standard of Care
Number analyzed (Participants) | 60 | 19
Hours | 8.85 (11.16) | 7.33 (4.51)
Statistical Analysis 1: Comparison: Cryoanalgesia + SOC vs Standard of Care; Analysis is the time from end of procedure to oral endotracheal extubation; Test type: Superiority; p = 0.4421, Wilcoxon (Mann-Whitney); Wilcoxon rank-sum test

7. Secondary Outcome: Secondary Outcome 5: Patient Controlled Analgesia (PCA) and Oral Opioid Consumption at the 24, 48, 96 and 120 Hour Time Points
Description: Patient Controlled Analgesia (PCA) is when the patient chooses to give themselves some form of analgesia, or painkiller, depending on their post-operation pain levels. Oral opioid consumption is the measure of all painkiller medicine that was prescribed by the hospital to the patient to take. This outcome measures each of these up to each time point and also measures the total PCA and oral opioid consumption post-procedure for the whole hospital stay.
Time Frame: 24-, 48, -96 and 120-hours
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalent (MME)
Arm/Group | Cryoanalgesia + SOC | Standard of Care
Number analyzed (Participants) | 63 | 19
Morphine Milligram Equivalent (MME)
  24 Hours | 11.43 (14.54) | 17.32 (23.65)
  48 Hours | 20.91 (23.45) | 31.05 (36.02)
  96 Hours: number analyzed (Participants) | 57 | 15
  96 Hours | 14.87 (19.82) | 16.67 (44.52)
  120 Hours: number analyzed (Participants) | 47 | 12
  120 Hours | 14.10 (18.58) | 13.13 (20.40)
  Total Post-Procedure for Hospital Stay | 33.43 (29.77) | 38.31 (31.05)
Statistical Analysis 1: Comparison: Cryoanalgesia + SOC vs Standard of Care; Test type: Superiority; p = 0.4352, Wilcoxon (Mann-Whitney) — Total Post-Procedure for Hospital Stay; Wilcoxon Rank-Sum Test

8. Secondary Outcome: Secondary Outcome 6: ICU and Hospital Length of Stay From Procedure to Discharge
Description: The outcome measures the time spent in the intensive care unit (ICU) as well as the total hospital length of stay.
Time Frame: Procedure to Discharge
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cryoanalgesia + SOC | Standard of Care
Number analyzed (Participants) | 60 | 19
Days
  ICU Length of Stay | 4.96 (7.75) | 2.96 (2.24)
  Hospital Length of Stay | 9.40 (8.34) | 6.32 (2.56)
Statistical Analysis 1: Comparison: Cryoanalgesia + SOC vs Standard of Care; Test type: Superiority; p = 0.2939, Wilcoxon (Mann-Whitney) — ICU Length of Stay; Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Cryoanalgesia + SOC vs Standard of Care; Test type: Superiority; p = 0.0998, Wilcoxon (Mann-Whitney) — Hospital Length of Stay; Wilcoxon rank-sum test

9. Secondary Outcome: Secondary Outcome 7: Ambulatory Movement During Hospital Stay
Description: Ambulatory Movement, defined as the subjects ability to sit up, stand up, walk and flex both the left and right shoulders, was measured at multiple time points during hospital stay.
Time Frame: Baseline, 48, 72, 96, 120 Hours and Discharge
Population: Initial patient population was 65 and 19 for the CRYO arm and SOC arm respectively. Number of patients analysed at the time points below differs due to the following: patient unwilling or refused test, patient discharged from hospital or other patient hospital stay issues.
Measure: Count of Participants; unit: Participants
Arm/Group | Cryoanalgesia + SOC | Standard of Care
Number analyzed (Participants) | 65 | 19
Participants
  Baseline - Able to sit up in bed: Yes - Independently | 65 | 19
  Baseline - Able to sit up in bed: Yes - with assistance | 0 | 0
  Baseline - Able to sit up in bed: No | 0 | 0
  Baseline - Able to stand up: Yes - Independently | 64 | 19
  Baseline - Able to stand up: Yes - with assistance | 1 | 0
  Baseline - Able to stand up: No | 0 | 0
  Baseline - Able to walk: Yes - Independently | 64 | 19
  Baseline - Able to walk: Yes - with assistance | 1 | 0
  Baseline - Able to walk: No | 0 | 0
  Baseline - Right shoulder flexion movement: Yes - Independently | 63 | 19
  Baseline - Right shoulder flexion movement: Yes - with assistance | 2 | 0
  Baseline - Right shoulder flexion movement: No | 0 | 0
  Baseline - Left shoulder flexion movement: Yes - Independently | 64 | 19
  Baseline - Left shoulder flexion movement: Yes - with assistance | 1 | 0
  Baseline - Left shoulder flexion movement: No | 0 | 0
  48 Hours - Able to sit up in bed: number analyzed (Participants) | 61 | 17
  48 Hours - Able to sit up in bed: Yes - Independently | 34 | 7
  48 Hours - Able to sit up in bed: Yes - with assistance | 27 | 10
  48 Hours - Able to sit up in bed: No | 0 | 0
  48 Hours - Able to stand up: number analyzed (Participants) | 61 | 17
  48 Hours - Able to stand up: Yes - Independently | 21 | 4
  48 Hours - Able to stand up: Yes - with assistance | 38 | 12
  48 Hours - Able to stand up: No | 2 | 1
  48 Hours - Able to walk: number analyzed (Participants) | 61 | 17
  48 Hours - Able to walk: Yes - Independently | 16 | 2
  48 Hours - Able to walk: Yes - with assistance | 38 | 13
  48 Hours - Able to walk: No | 7 | 2
  48 Hours - Right shoulder flexion movement: number analyzed (Participants) | 61 | 16
  48 Hours - Right shoulder flexion movement: Yes - Independently | 26 | 8
  48 Hours - Right shoulder flexion movement: Yes - with assistance | 33 | 8
  48 Hours - Right shoulder flexion movement: No | 2 | 0
  48 Hours - Left shoulder flexion movement: number analyzed (Participants) | 61 | 16
  48 Hours - Left shoulder flexion movement: Yes - Independently | 43 | 12
  48 Hours - Left shoulder flexion movement: Yes - with assistance | 16 | 4
  48 Hours - Left shoulder flexion movement: No | 2 | 0
  72 Hours - Able to sit up in bed: number analyzed (Participants) | 59 | 17
  72 Hours - Able to sit up in bed: Yes - Independently | 47 | 8
  72 Hours - Able to sit up in bed: Yes - with assistance | 12 | 9
  72 Hours - Able to sit up in bed: No | 0 | 0
  72 Hours - Able to stand up: number analyzed (Participants) | 59 | 17
  72 Hours - Able to stand up: Yes - Independently | 39 | 5
  72 Hours - Able to stand up: Yes - with assistance | 20 | 10
  72 Hours - Able to stand up: No | 0 | 2
  72 Hours - Able to walk: number analyzed (Participants) | 59 | 17
  72 Hours - Able to walk: Yes - Independently | 28 | 4
  72 Hours - Able to walk: Yes - with assistance | 27 | 11
  72 Hours - Able to walk: No | 4 | 2
  72 Hours - Right shoulder flexion movement: number analyzed (Participants) | 59 | 17
  72 Hours - Right shoulder flexion movement: Yes - Independently | 41 | 12
  72 Hours - Right shoulder flexion movement: Yes - with assistance | 17 | 5
  72 Hours - Right shoulder flexion movement: No | 1 | 0
  72 Hours - Left shoulder flexion movement: number analyzed (Participants) | 59 | 17
  72 Hours - Left shoulder flexion movement: Yes - Independently | 49 | 15
  72 Hours - Left shoulder flexion movement: Yes - with assistance | 8 | 2
  72 Hours - Left shoulder flexion movement: No | 2 | 0
  96 Hours - Able to sit up in bed: number analyzed (Participants) | 51 | 15
  96 Hours - Able to sit up in bed: Yes - Independently | 41 | 12
  96 Hours - Able to sit up in bed: Yes - with assistance | 10 | 3
  96 Hours - Able to sit up in bed: No | 0 | 0
  96 Hours - Able to stand up: number analyzed (Participants) | 51 | 15
  96 Hours - Able to stand up: Yes - Independently | 32 | 8
  96 Hours - Able to stand up: Yes - with assistance | 19 | 6
  96 Hours - Able to stand up: No | 0 | 1
  96 Hours - Able to walk: number analyzed (Participants) | 51 | 15
  96 Hours - Able to walk: Yes - Independently | 26 | 7
  96 Hours - Able to walk: Yes - with assistance | 21 | 7
  96 Hours - Able to walk: No | 4 | 1
  96 Hours - Right shoulder flexion movement: number analyzed (Participants) | 51 | 15
  96 Hours - Right shoulder flexion movement: Yes - Independently | 39 | 11
  96 Hours - Right shoulder flexion movement: Yes - with assistance | 11 | 4
  96 Hours - Right shoulder flexion movement: No | 1 | 0
  96 Hours - Left shoulder flexion movement: number analyzed (Participants) | 51 | 15
  96 Hours - Left shoulder flexion movement: Yes - Independently | 43 | 13
  96 Hours - Left shoulder flexion movement: Yes - with assistance | 6 | 2
  96 Hours - Left shoulder flexion movement: No | 2 | 0
  120 Hours - Able to sit up in bed: number analyzed (Participants) | 42 | 10
  120 Hours - Able to sit up in bed: Yes - Independently | 36 | 7
  120 Hours - Able to sit up in bed: Yes - with assistance | 6 | 3
  120 Hours - Able to sit up in bed: No | 0 | 0
  120 Hours - Able to stand up: number analyzed (Participants) | 42 | 10
  120 Hours - Able to stand up: Yes - Independently | 30 | 5
  120 Hours - Able to stand up: Yes - with assistance | 12 | 5
  120 Hours - Able to stand up: No | 0 | 0
  120 Hours - Able to walk: number analyzed (Participants) | 42 | 10
  120 Hours - Able to walk: Yes - Independently | 23 | 5
  120 Hours - Able to walk: Yes - with assistance | 17 | 5
  120 Hours - Able to walk: No | 2 | 0
  120 Hours - Right shoulder flexion movement: number analyzed (Participants) | 42 | 10
  120 Hours - Right shoulder flexion movement: Yes - Independently | 34 | 9
  120 Hours - Right shoulder flexion movement: Yes - with assistance | 8 | 1
  120 Hours - Right shoulder flexion movement: No | 0 | 0
  120 Hours - Left shoulder flexion movement: number analyzed (Participants) | 42 | 10
  120 Hours - Left shoulder flexion movement: Yes - Independently | 37 | 10
  120 Hours - Left shoulder flexion movement: Yes - with assistance | 5 | 0
  120 Hours - Left shoulder flexion movement: No | 0 | 0
  Discharge - Able to sit up in bed: number analyzed (Participants) | 60 | 19
  Discharge - Able to sit up in bed: Yes - Independently | 53 | 19
  Discharge - Able to sit up in bed: Yes - with assistance | 7 | 0
  Discharge - Able to sit up in bed: No | 0 | 0
  Discharge - Able to stand up: number analyzed (Participants) | 60 | 19
  Discharge - Able to stand up: Yes - Independently | 51 | 17
  Discharge - Able to stand up: Yes - with assistance | 7 | 2
  Discharge - Able to stand up: No | 2 | 0
  Discharge - Able to walk: number analyzed (Participants) | 60 | 19
  Discharge - Able to walk: Yes - Independently | 50 | 15
  Discharge - Able to walk: Yes - with assistance | 8 | 4
  Discharge - Able to walk: No | 2 | 0
  Discharge - Right shoulder flexion movement: number analyzed (Participants) | 60 | 19
  Discharge - Right shoulder flexion movement: Yes - Independently | 54 | 16
  Discharge - Right shoulder flexion movement: Yes - with assistance | 6 | 3
  Discharge - Right shoulder flexion movement: No | 0 | 0
  Discharge - Left shoulder flexion movement: number analyzed (Participants) | 60 | 19
  Discharge - Left shoulder flexion movement: Yes - Independently | 51 | 16
  Discharge - Left shoulder flexion movement: Yes - with assistance | 5 | 3
  Discharge - Left shoulder flexion movement: No | 4 | 0
Statistical Analysis 1: Comparison: Cryoanalgesia + SOC vs Standard of Care; 48 Hours Post-Op: Patient able to sit up in bed; Test type: Superiority; p = 0.2877, Chi-squared
Statistical Analysis 2: Comparison: Cryoanalgesia + SOC vs Standard of Care; 48 Hours Post-Op: Patient able to stand up; Test type: Superiority; p = 0.5311, Fisher Exact
Statistical Analysis 3: Comparison: Cryoanalgesia + SOC vs Standard of Care; 48 Hours Post-Op: Patient able to walk; Test type: Superiority; p = 0.4908, Fisher Exact
Statistical Analysis 4: Comparison: Cryoanalgesia + SOC vs Standard of Care; 48 Hours Post-Op: Right Shoulder Flexion Movement; Test type: Superiority; p = 0.8621, Fisher Exact
Statistical Analysis 5: Comparison: Cryoanalgesia + SOC vs Standard of Care; 48 Hours Post-Op: Left Shoulder Flexion Movement; Test type: Superiority; p = 1, Fisher Exact
Statistical Analysis 6: Comparison: Cryoanalgesia + SOC vs Standard of Care; 72 Hours Post-Op: Patient able to sit up in bed; Test type: Superiority; p = 0.0133, Fisher Exact
Statistical Analysis 7: Comparison: Cryoanalgesia + SOC vs Standard of Care; 72 Hours Post-Op: Patient able to stand up; Test type: Superiority; p = 0.0037, Fisher Exact
Statistical Analysis 8: Comparison: Cryoanalgesia + SOC vs Standard of Care; 72 Hours Post-Op: Patient able to walk; Test type: Superiority; p = 0.1671, Fisher Exact
Statistical Analysis 9: Comparison: Cryoanalgesia + SOC vs Standard of Care; 72 Hours Post-Op: Right Shoulder Flexion Movement; Test type: Superiority; p = 1.000, Fisher Exact
Statistical Analysis 10: Comparison: Cryoanalgesia + SOC vs Standard of Care; 72 Hours Post-Op: Left Shoulder Flexion Movement; Test type: Superiority; p = 1, Fisher Exact
Statistical Analysis 11: Comparison: Cryoanalgesia + SOC vs Standard of Care; 96 Hours Post-Op: Patient able to sit up in bed; Test type: Superiority; p = 1, Fisher Exact
Statistical Analysis 12: Comparison: Cryoanalgesia + SOC vs Standard of Care; 96 Hours Post-Op: Patient able to stand up; Test type: Superiority; p = 0.2757, Fisher Exact
Statistical Analysis 13: Comparison: Cryoanalgesia + SOC vs Standard of Care; 96 Hours Post-Op: Patient able to walk; Test type: Superiority; p = 0.9025, Fisher Exact
Statistical Analysis 14: Comparison: Cryoanalgesia + SOC vs Standard of Care; 96 Hours Post-Op: Right Shoulder Flexion Movement; Test type: Superiority; p = 0.7942, Fisher Exact
Statistical Analysis 15: Comparison: Cryoanalgesia + SOC vs Standard of Care; 96 Hours Post-Op: Left Shoulder Flexion Movement; Test type: Superiority; p = 1, Fisher Exact
Statistical Analysis 16: Comparison: Cryoanalgesia + SOC vs Standard of Care; 120 Hours Post-Op: Patient able to sit up in bed; Test type: Superiority; p = 0.3492, Fisher Exact
Statistical Analysis 17: Comparison: Cryoanalgesia + SOC vs Standard of Care; 120 Hours Post-Op: Patient able to stand up; Test type: Superiority; p = 0.2644, Fisher Exact
Statistical Analysis 18: Comparison: Cryoanalgesia + SOC vs Standard of Care; 120 Hours Post-Op: Patient able to walk; Test type: Superiority; p = 0.8258, Fisher Exact
Statistical Analysis 19: Comparison: Cryoanalgesia + SOC vs Standard of Care; 120 Hours Post-Op: Right Shoulder Flexion Movement; Test type: Superiority; p = 0.67, Fisher Exact
Statistical Analysis 20: Comparison: Cryoanalgesia + SOC vs Standard of Care; 120 Hours Post-Op: Left Shoulder Flexion Movement; Test type: Superiority; p = 0.5693, Fisher Exact
Statistical Analysis 21: Comparison: Cryoanalgesia + SOC vs Standard of Care; Discharge: Patient able to sit up in bed; Test type: Superiority; p = 0.1189, Chi-squared
Statistical Analysis 22: Comparison: Cryoanalgesia + SOC vs Standard of Care; Discharge: Patient able to stand up; Test type: Superiority; p = 1, Fisher Exact
Statistical Analysis 23: Comparison: Cryoanalgesia + SOC vs Standard of Care; Discharge: Patient able to walk; Test type: Superiority; p = 0.6992, Fisher Exact
Statistical Analysis 24: Comparison: Cryoanalgesia + SOC vs Standard of Care; Discharge: Right Shoulder Flexion Movement; Test type: Superiority; p = 0.4429, Fisher Exact
Statistical Analysis 25: Comparison: Cryoanalgesia + SOC vs Standard of Care; Discharge: Left Shoulder Flexion Movement; Test type: Superiority; p = 0.4563, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse event data was captured over the entirety of the study, starting at the Baseline Visit and ending at the 6 Month Visit, which was the study exit visit.
Description: The Investigator at each participating site was responsible for reporting Adverse Events (AEs) and Serious Adverse Events (SAEs) to AtriCure only when they were related to the CryoAnalgesia index procedure or device, therefore access to all adverse events is not possible. All AEs reported to AtriCure (i.e., AEs related to the CryoAnalgesia procedure or device) will be reported.
Arm/Group | Cryoanalgesia + SOC | Standard of Care
All-Cause Mortality (participants affected / at risk) | 8/65 | 1/19
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/19
Other Adverse Events (participants affected / at risk) | 2/65 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryoanalgesia + SOC (N=65) | Standard of Care (N=19)
Right Breast Pain/Numbness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyperesthesia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-09-26): https://cdn.clinicaltrials.gov/large-docs/53/NCT02922153/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT02922153/Prot_SAP_001.pdf